CLINICAL TRIAL: NCT03597087
Title: The Difference of Two Year Recurrence Rate According to Anesthetic Method During Transurethral Resection of Bladder Mass in Patients With Non-muscle Invasive Bladder Cancer: Prospective, Randomized, Clinical Phase II Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ja Hyeon Ku, Professor, MD., PHD., Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SeoulNUH_2018_TURBT
Record Dates: First submitted 2018-07-02; First posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Bladder Cancer
Keywords: Anesthesia, Bladder cancer, Recurrence rate, Transurethral resection of bladder mass
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Anesthesia

STUDY DESIGN:
Intervention Model Description: After randomization, they were divided into two parallel groups 289 patients were randomly assigned to a spinal anesthesia group and a general anesthesia group 1: 1.
Masking Description: Using a web site, and creating a randomized list at Sealedenvalop.com. Patients are randomly assigned to receive an anesthetic consent, and no masking is performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia (Experimental): Group of general anesthesia before transurethral resection of the bladder tumor anesthesia: propopol
  Interventions: Procedure: Anesthesia before transurethral resection of the bladder tumor; Drug: Anesthesia
- Spinal anesthesia (Experimental): Group of spinal anesthesia before transurethral resection of the bladder tumor anesthesia: bupibacaine
  Interventions: Procedure: Anesthesia before transurethral resection of the bladder tumor; Drug: Anesthesia

INTERVENTIONS:
Procedure: Anesthesia before transurethral resection of the bladder tumor — General anaesthesia or general anesthesia (see spelling differences) is a medically induced coma with loss of protective reflexes, resulting from the administration of one or more general anaesthetic agents.
  Spinal anaesthesia is a form of regional anaesthesia involving the injection of a local anaesthetic into the subarachnoid space, generally through a fine needle
Drug: Anesthesia — General anaesthesia : propopol
  Spinal anaesthesia : bupibacaine

SUMMARY:
The investigators compare the recurrence rate difference between two years after transurethral resection of the bladder tumor according to the method of anesthesia. Anesthetic methods are general anesthesia and spinal anesthesia. Assessment of recurrence is assessed by bladder endoscopy, CT, and pathological examination of surgical specimens.

DETAILED DESCRIPTION:
1. Research Background Most of the bladder cancer (approximately 85%) has histologic features of urothelial carcinoma. Approximately 75% of the patients initially diagnosed as non-invasive bladder cancer (stage I, CIS) or submucosal stage T1 -muscle invasive bladder cancer - NMIBC). However, it has been reported that about 60% to 70% of patients experience recurrence and 20% to 30% of relapsed cancers require radical cystectomy or chemotherapy It is known to progress to high-grade or high grade cancer.

   There are studies that involve surgical factors such as volatile anesthetics, narcotic analgesics, anti-body temperature, blood transfusion, and cancer recurrence. Minimizing the use of volatile anesthetics and narcotic analgesics reduces spinal anesthesia before and after surgery, It has been reported that there is a correlation with maintenance of immune cell function
2. Research hypothesis and purpose The aim of this study was to evaluate the recurrence rate, recurrence - free survival rate, and recurrence - free survival rate of non - muscle invasive bladder carcinoma in patients undergoing bladder resection.
3. Research Method

   * Preoperative screening: Physical examination, Blood test, CT urography, Urine analysis, Urine culture, Urine cytology, Cystoscopy. Enforced
   * Randomization on the day before surgery: 289 patients were randomly assigned to a spinal anesthesia group and a general anesthesia group 1: 1.

Urine analysis, urine culture, urine cytology, and cystoscopy were performed every 3 months up to 2 years postoperatively. CT urography performed once a year

* Follow-up procedure: Follow-up procedure according to bladder cancer standard.

  4. Observation items, clinical examination items and observational examination methods
* Screening: CT urography, Urine analysis, Urine culture, Urine cytology, Cystoscopy. Observe
* Follow up: Urine analysis, Urine culture, Urine cytology, Cystoscopy every 3 months after the operation, CT urography every year

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older
2. Patients with suspected Ta / T1 non-muscle invasive bladder cancer
3. Patients who were not previously treated with other cancers
4. Normal range creatinine, AST, ALT patients
5. Patients with both spinal anesthesia and general anesthesia

Exclusion Criteria:

1. Patients with urinary tract carcinoma not invading the renal pelvis, ureter or urethra
2. Patients with cancer other than bladder cancer or a history of treatment
3. Patients with clinical evidence of muscle-invasive bladder cancer
4. Patients taking immunosuppressive drugs and immunosuppressive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 289 (Estimated)
Dates: Start 2018-07-19 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence-free survival rate | Follow up every 3 months until 2 years after surgery
  The criteria for recurrence-free survival and recurrence of bladder cancer for 2 years postoperatively are based on pathological histology. If the recurrence is suspected in the radiological examination but pathological histological examination is difficult, the reference is based on the day of the imaging examination suspected of recurrence.

SECONDARY OUTCOMES:
2-year progression-free survival | Follow up every 3 months until 2 years after surgery
  The progression-free survival rate and progression rate of bladder cancer for 2 years postoperatively include both T stage and tumor grade progression.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Tae Kim, PhD, Study Director — Professor, Department of Anesthesiology, Seoul National University Hospital; Ja Hyeon Ku, PhD, Study Chair — Professor, Department of Urology, Seoul National University Hospital; Hyeong Dong Yuk, MD, Principal Investigator — Clinical fellow, Department of Urology, Seoul National University Hospital; Song Hee Kim, Bacheolor, Principal Investigator — Researcher, Department of Urology, Seoul National University Hospital; Jae Hyun Jung, MD, Principal Investigator — Clinical fellow, Department of Urology, Seoul National University Hospital; Jung Hoon Lee, MD, Principal Investigator — Clinical fellow, Department of Urology, Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Herr HW, Faulkner JR, Grossman HB, Natale RB, deVere White R, Sarosdy MF, Crawford ED. Surgical factors influence bladder cancer outcomes: a cooperative group report. J Clin Oncol. 2004 Jul 15;22(14):2781-9. doi: 10.1200/JCO.2004.11.024. Epub 2004 Jun 15. PMID 15199091
- [Result] Christodouleas JP, Baumann BC, He J, Hwang WT, Tucker KN, Bekelman JE, Tangen CM, Lerner SP, Guzzo TJ, Malkowicz SB, Herr H. Optimizing bladder cancer locoregional failure risk stratification after radical cystectomy using SWOG 8710. Cancer. 2014 Apr 15;120(8):1272-80. doi: 10.1002/cncr.28544. Epub 2014 Jan 3. PMID 24390799
- [Result] Witjes JA, Comperat E, Cowan NC, De Santis M, Gakis G, Lebret T, Ribal MJ, Van der Heijden AG, Sherif A; European Association of Urology. EAU guidelines on muscle-invasive and metastatic bladder cancer: summary of the 2013 guidelines. Eur Urol. 2014 Apr;65(4):778-92. doi: 10.1016/j.eururo.2013.11.046. Epub 2013 Dec 12. PMID 24373477
- [Result] Pollack A, Zagars GK, Cole CJ, Dinney CP, Swanson DA, Grossman HB. The relationship of local control to distant metastasis in muscle invasive bladder cancer. J Urol. 1995 Dec;154(6):2059-63; discussion 2063-4. PMID 7500458
- [Result] Jensen JB, Ulhoi BP, Jensen KM. Extended versus limited lymph node dissection in radical cystectomy: impact on recurrence pattern and survival. Int J Urol. 2012 Jan;19(1):39-47. doi: 10.1111/j.1442-2042.2011.02887.x. Epub 2011 Nov 3. PMID 22050425
- [Result] Zaghloul MS, Awwad HK, Akoush HH, Omar S, Soliman O, el Attar I. Postoperative radiotherapy of carcinoma in bilharzial bladder: improved disease free survival through improving local control. Int J Radiat Oncol Biol Phys. 1992;23(3):511-7. doi: 10.1016/0360-3016(92)90005-3. PMID 1612951
- [Result] Lawton CA, Michalski J, El-Naqa I, Buyyounouski MK, Lee WR, Menard C, O'Meara E, Rosenthal SA, Ritter M, Seider M. RTOG GU Radiation oncology specialists reach consensus on pelvic lymph node volumes for high-risk prostate cancer. Int J Radiat Oncol Biol Phys. 2009 Jun 1;74(2):383-7. doi: 10.1016/j.ijrobp.2008.08.002. Epub 2008 Oct 22. PMID 18947938
- [Result] Baumann BC, Guzzo TJ, He J, Keefe SM, Tucker K, Bekelman JE, Hwang WT, Vaughn DJ, Malkowicz SB, Christodouleas JP. A novel risk stratification to predict local-regional failures in urothelial carcinoma of the bladder after radical cystectomy. Int J Radiat Oncol Biol Phys. 2013 Jan 1;85(1):81-8. doi: 10.1016/j.ijrobp.2012.03.007. Epub 2012 Apr 28. PMID 22543204
- [Result] Baumann BC, Guzzo TJ, He J, Vaughn DJ, Keefe SM, Vapiwala N, Deville C, Bekelman JE, Tucker K, Hwang WT, Malkowicz SB, Christodouleas JP. Bladder cancer patterns of pelvic failure: implications for adjuvant radiation therapy. Int J Radiat Oncol Biol Phys. 2013 Feb 1;85(2):363-9. doi: 10.1016/j.ijrobp.2012.03.061. Epub 2012 May 30. PMID 22658217
- [Result] Ku JH, Kim M, Jeong CW, Kwak C, Kim HH. Risk prediction models of locoregional failure after radical cystectomy for urothelial carcinoma: external validation in a cohort of korean patients. Int J Radiat Oncol Biol Phys. 2014 Aug 1;89(5):1032-1037. doi: 10.1016/j.ijrobp.2014.04.049. Epub 2014 Jul 8. PMID 25035206
- [Result] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Result] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Result] Babjuk M, Burger M, Comperat E, Palou J, Roupret M, van Rhijn B, Shariat S, Sylvester R, Zigeuner R, Gontero P, Mostafid H. Reply to Harry Herr's Letter to the Editor re: Marko Babjuk, Andreas Bohle, Maximilian Burger, et al. EAU Guidelines on Non-muscle-invasive Urothelial Carcinoma of the Bladder: Update 2016. Eur Urol 2017;71:447-61. Eur Urol. 2017 Jun;71(6):e173-e174. doi: 10.1016/j.eururo.2016.11.029. Epub 2016 Dec 7. No abstract available. PMID 27939074
- [Result] Burger M, Catto JW, Dalbagni G, Grossman HB, Herr H, Karakiewicz P, Kassouf W, Kiemeney LA, La Vecchia C, Shariat S, Lotan Y. Epidemiology and risk factors of urothelial bladder cancer. Eur Urol. 2013 Feb;63(2):234-41. doi: 10.1016/j.eururo.2012.07.033. Epub 2012 Jul 25. PMID 22877502
- [Result] Kamat AM, Witjes JA, Brausi M, Soloway M, Lamm D, Persad R, Buckley R, Bohle A, Colombel M, Palou J. Defining and treating the spectrum of intermediate risk nonmuscle invasive bladder cancer. J Urol. 2014 Aug;192(2):305-15. doi: 10.1016/j.juro.2014.02.2573. Epub 2014 Mar 25. PMID 24681333
- [Result] Hall MC, Chang SS, Dalbagni G, Pruthi RS, Seigne JD, Skinner EC, Wolf JS Jr, Schellhammer PF. Guideline for the management of nonmuscle invasive bladder cancer (stages Ta, T1, and Tis): 2007 update. J Urol. 2007 Dec;178(6):2314-30. doi: 10.1016/j.juro.2007.09.003. No abstract available. PMID 17993339
- [Result] Morales A, Eidinger D, Bruce AW. Intracavitary Bacillus Calmette-Guerin in the treatment of superficial bladder tumors. J Urol. 1976 Aug;116(2):180-3. doi: 10.1016/s0022-5347(17)58737-6. PMID 820877
- [Result] Balkwill F, Mantovani A. Inflammation and cancer: back to Virchow? Lancet. 2001 Feb 17;357(9255):539-45. doi: 10.1016/S0140-6736(00)04046-0. PMID 11229684
- [Result] Grivennikov SI, Greten FR, Karin M. Immunity, inflammation, and cancer. Cell. 2010 Mar 19;140(6):883-99. doi: 10.1016/j.cell.2010.01.025. PMID 20303878
- [Result] Kim HS, Ku JH. Systemic Inflammatory Response Based on Neutrophil-to-Lymphocyte Ratio as a Prognostic Marker in Bladder Cancer. Dis Markers. 2016;2016:8345286. doi: 10.1155/2016/8345286. Epub 2016 Jan 5. PMID 26880857
- [Result] Crumley AB, McMillan DC, McKernan M, Going JJ, Shearer CJ, Stuart RC. An elevated C-reactive protein concentration, prior to surgery, predicts poor cancer-specific survival in patients undergoing resection for gastro-oesophageal cancer. Br J Cancer. 2006 Jun 5;94(11):1568-71. doi: 10.1038/sj.bjc.6603150. PMID 16685271
- [Result] Dutta S, Crumley AB, Fullarton GM, Horgan PG, McMillan DC. Comparison of the prognostic value of tumour and patient related factors in patients undergoing potentially curative resection of gastric cancer. Am J Surg. 2012 Sep;204(3):294-9. doi: 10.1016/j.amjsurg.2011.10.015. Epub 2012 Mar 22. PMID 22444831
- [Result] Kweon TD, Lee KY. Spinal anesthesia is associated with lower recurrence rates after resection of non-muscle invasive bladder cancer. Transl Androl Urol. 2018 Apr;7(2):283-286. doi: 10.21037/tau.2018.03.13. No abstract available. PMID 29733090
- [Derived] Han JH, Yuk HD, Jeong SH, Jeong CW, Kwak C, Kim JT, Ku JH. Anesthetic approaches and 2-year recurrence rates in non-muscle invasive bladder cancer: a randomized clinical trial. Reg Anesth Pain Med. 2024 Dec 31:rapm-2024-105949. doi: 10.1136/rapm-2024-105949. Online ahead of print. PMID 39740955